CLINICAL TRIAL: NCT00235326
Title: Chronic Gastrointestinal Sequelae of an Acute Outbreak of Bacterial Gastroenteritis in Walkerton Ontario
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: John Marshall, Mcmaster University
Other Study IDs: 02-026; 05-346
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: residents of Walkerton ontario at outbreak
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Unexposed to gastroenteritis
- 1: Exposed to gastroenteritis

SUMMARY:
Acute Bacterial dysentery leads to chronic symptoms of disturbed bowel habit in a minority of individuals. This condition known as post infectious irritable bowel syndrome (PI-IBS) remains poorly understood. This could allow material in the bowel to reach deeper tissues of the bowel wall leading to inflammation and changes in muscle and nerve function. This is also early evidence that genetic programming of people with PI-IBS prevents them from turning off inflammation once it begins. Literature suggests that IBS may develop at greater rates in individuals with pro-inflammatory genotype and that these individuals may be at increased risk of inflammatory bowel diseases (IBD).

DETAILED DESCRIPTION:
This research will study chronic gastrointestinal problems in the residents of Walkerton, Ontario region. Determine whether acute bacterial infection is a risk factor for development of inflammatory bowel disease using the population of Walkerton as a cohort. We hypothesize that exposure to bacterial infection leads to development of post infectious irritable bowel syndrome which is associated with an increase in intestinal permeability and immune activation with low grade intestinal inflammation and that this sequence of events will trigger inflammatory bowel disease in genetically susceptible individuals

ELIGIBILITY:
Inclusion Criteria:

* Participants must be residents of the Walkerton, Ontario region at the time of Outbreak who consented to the study

Exclusion Criteria:

* Non residents of Walkerton Ontario at the time of outbreak

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: residents of walkerton
Sampling Method: Non-Probability Sample
Enrollment: 4561 (Actual)
Dates: Start 2002-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John k Marshall, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- Walkerton, Walkerton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Residents of Walkerton in may 2000
Pre-assignment Details: Age less than 16, non-residents of walkerton, premorbid Inflammatory Bowel disease(IBD) /Irritable bowel syndrome(IBS)
Period: Overall Study
Arm/Group | Unexposed to Gastroenteritis | Exposed to Gastroenteritis
Started | 1575 | 2986
Completed | 829 | 1586
Not Completed | 746 | 1400
Not completed — Lost to Follow-up | 746 | 1400

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unexposed to Gastroenteritis | Exposed to Gastroenteritis | Total
Number analyzed (Participants) | 1575 | 2986 | 4561
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 471 | 907 | 1378.0
  Between 18 and 65 years | 905 | 1810 | 2715.0
  >=65 years | 199 | 269 | 468.0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.96 (22.76) | 34.97 (21.61) | 35.66 (22.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 892 | 1665 | 2557.0
  Male | 683 | 1321 | 2004.0
Region of Enrollment [Number; unit: participants]
  Canada | 1575 | 2986 | 4561.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post Infectious Irritable Bowel Syndrome
Time Frame: 8 years
Measure: Number; unit: participants
Arm/Group | Unexposed to Gastroenteritis | Exposed to Gastroenteritis
Number analyzed (Participants) | 829 | 1586
participants | 23 | 114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less